CLINICAL TRIAL: NCT05215262
Title: TAKE Steps: Motivational Interviewing to Improve Comprehensive HIV and Sexually Transmitted Infection Prevention in Adolescent Primary Care
Brief Title: TAKE Steps: Motivational Interviewing to Prevent STIs
Acronym: TAKE Steps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-016708; K23MH119976-02 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Self Efficacy; HIV Prevention; STI Prevention
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T.A.K.E. Steps Motivational Interviewing Intervention (Experimental): Four MI intervention sessions, 1:1 with participant and health coach.
  Interventions: Behavioral: Treat Act Know Engage (T.A.K.E.) Steps
- Standard of Care (Active Comparator): Standard of Care control visit with primary care physician (PCP)
  Interventions: Behavioral: Standard or Care

INTERVENTIONS:
Behavioral: Treat Act Know Engage (T.A.K.E.) Steps — Intervention sessions will consist of psychoeducation, HIV/STI goal identification, referral to HIV testing and PrEP, and communication skill building.
  Arms: T.A.K.E. Steps Motivational Interviewing Intervention
Behavioral: Standard or Care — S.O.C. arm will receive treatment as usual. After the baseline interview, participants will be referred to their PCP for management of any clinical issues that arise. Their clinic visit schedule will follow their clinical needs and recommendations of their clinic provider
  Arms: Standard of Care

SUMMARY:
This study will consist of a randomized controlled trial of a motivational interviewing intervention for adolescents with diagnosed sexually transmitted infections (STIs). The sessions will provide HIV/STI prevention education, use motivational interviewing (MI) to enhance goal setting, and providing skill building and referral to evidence based STI and HIV prevention strategies Pre-Exposure Prophylaxis (PrEP), condom use, and partner notification.

DETAILED DESCRIPTION:
Pilot phase: Pilot testing will occur over a 3-month period to prime intervention for implementation, with the aim of recruiting n=10 pilot participants. Pilot phase participants will follow the same study procedure timeline as participants randomized to the MI intervention arm of the randomized control trial (RCT), excluding the 6-month follow-up visit. Pilot participants will not be followed in the RCT or contribute outcome data. At the end of every intervention visit in the pilot phase (the baseline, 1-week, 1-month and 3-month visits), participants will complete a brief feedback interview to ensure face validity and identify areas needing refinement. Feedback will be incorporated into the study design, with amendments submitted to the Institutional Review Board (IRB) as needed. Data from pilot participants will not be included in analysis of the RCT.

Intervention phase:The RCT will randomize youth with recent STI 2:1 to the TAKE Steps intervention vs a standard of care (SOC) control. Both arms (intervention and SOC) will have data collection visits at the baseline, the 3-month, and the 6-month-follow-up time points. In addition, the intervention group will have intervention sessions at baseline, 1 week, 1 month and 3 months.

The study treatment phase for the RCT will consist of data collection and motivational interviewing sessions over a 6-month period. Intervention sessions will consist of HIV and STI prevention education, motivational interviewing, skill building, and referral to therapy.

All visits can occur in-person or remotely.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 13 to 19 years.
* History of ≥1 STI in the 30 days prior to recruitment
* Confirmed treatment for a laboratory confirmed diagnosis of Trichomonas vaginalis (via microscopy or nucleic acid amplification test [NAAT]), Neisseria gonorrhea (NAAT), Chlamydia trachomatis (NAAT), Treponema pallidum [via new positive rapid plasmin reagin (RPR) assay] within the prior 30 days
* Self-reported HIV negative status.
* Able to speak and understand written English

Exclusion Criteria:

* Unable to provide informed consent due to intoxication or severe psychological distress.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Wood, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Primary Care, CHOP Clinic 3550 Market St, Philadelphia, Pennsylvania
  - CHOP Primary Care, Roxborough, Philadelphia, Pennsylvania
  - CHOP Karabots Pediatric Care Center, West Philadelphia, Philadelphia, Pennsylvania
  - CHOP Primary Care, Cobbs Creek, Philadelphia, Pennsylvania
  - CHOP Primary Care, South Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T.A.K.E. Steps Motivational Interviewing Intervention | Standard of Care
Started | 54 | 40
Completed | 42 | 40
Not Completed | 12 | 0
Not completed — Lost to Follow-up | 12 | 0

BASELINE CHARACTERISTICS:
Population: Only 42 of the 54 allocated to the intervention had Baseline data used for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | T.A.K.E. Steps Motivational Interviewing Intervention | Standard of Care | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only 42 of the 54 allocated to the intervention had Baseline data used for analysis.
  years | 16.6 (1) | 17.0 (1) | 16.8 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 37 | 32 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 37 | 75
  White | 1 | 0 | 1
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Prevention Self-efficacy
Description: Differences in the change in prevention self-efficacy scores from baseline to three months between the control arm compared to the intervention arm will be assessed using a modified version of the Generalized Self Efficacy (GSE) measure. The GSE measure is a 10-item measure assessing participants' confidence in carrying out their self-identified prevention goals. The total score of the GSE measure is calculated by finding the sum of all 10 items - the sum ranging between 10 and 40 with a higher score indicating more self-efficacy. This outcome is measuring the differences in mean total scores over time.
Time Frame: Baseline and 3 months
Population: Change in prevention self-efficacy score from Baseline to Three Months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | T.A.K.E. Steps Motivational Interviewing Intervention | Standard of Care
Number analyzed (Participants) | 42 | 40
score on a scale | 1.87 [0.04 to 3.17] | 0.20 [-1.59 to 1.99]
Statistical Analysis 1: Comparison: T.A.K.E. Steps Motivational Interviewing Intervention; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 1.87, 95% CI 2-sided [0.04 to 3.17]
Statistical Analysis 2: Comparison: Standard of Care; Test type: Superiority; p = 0.82, Mixed Models Analysis; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-1.59 to 1.99]
Statistical Analysis 3: Comparison: T.A.K.E. Steps Motivational Interviewing Intervention vs Standard of Care; Difference-in-differences results, comparing GSES scores between the Intervention and Standard of Care groups at the three-month time point; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [-0.89 to 4.23]

2. Secondary Outcome: Recruitment Feasibility
Description: Feasibility of recruitment will be measured by calculating the proportion of patients enrolled / patients recruited.
Time Frame: Baseline
Population: Total number of patients recruited.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Enrolled/Recruited: Patients recruited for study participation.
Arm/Group | Patients Enrolled/Recruited
Number analyzed (Participants) | 639
Participants | 94

3. Secondary Outcome: Intervention Acceptability
Description: Intervention acceptability will be measured at 1-week and 3-months by a 7-item satisfaction survey. This outcome measures the percentage participants who agreed or strongly agreed with statements on a 7-item acceptability survey completed at their 1-week intervention coaching session.
Time Frame: 1 week
Population: This analysis is based on a sample size of n=26 intervention participants who completed acceptability surveys at their 1-week intervention coaching sessions. Surveys asked participants for their agreement level of satisfaction on 7 statements about the intervention sessions. All 26 participants showed agreement or strong agreement with the 7 statements.
Measure: Count of Participants; unit: Participants
Groups:
- Participant Percentage of Agreement and Strong Agreement With Acceptability Statements: Four MI intervention sessions, 1:1 with participant and health coach.
  Treat Act Know Engage (T.A.K.E.) Steps: Intervention sessions will consist of psychoeducation, HIV/STI goal identification, referral to HIV testing and PrEP, and communication skill building.
  This group completed their 1-week coaching session and completed a 1-week acceptability survey.
Arm/Group | Participant Percentage of Agreement and Strong Agreement With Acceptability Statements
Number analyzed (Participants) | 26
Participants | 26

4. Secondary Outcome: Intervention Acceptability
Description: Intervention acceptability will be measured at 1-week and 3-months by a 7-item satisfaction survey. This outcome measures the percentage participants who agreed or strongly agreed with statements on a 7-item acceptability survey completed at their 3-month intervention coaching session.
Time Frame: 3 months
Population: This analysis is based on a sample size of n=27 intervention participants who completed acceptability surveys at their 3-month intervention coaching sessions. Surveys asked participants for their agreement level of satisfaction on 7 statements about the intervention sessions. All 27 participants showed agreement or strong agreement with the 7 statements.
Measure: Count of Participants; unit: Participants
Groups:
- Participant Percentage of Agreement and Strong Agreement With Acceptability Statements: Four MI intervention sessions, 1:1 with participant and health coach.
  Treat Act Know Engage (T.A.K.E.) Steps: Intervention sessions will consist of psychoeducation, HIV/STI goal identification, referral to HIV testing and PrEP, and communication skill building.
  This group completed their 3-month coaching session and completed a 3-month acceptability survey.
Arm/Group | Participant Percentage of Agreement and Strong Agreement With Acceptability Statements
Number analyzed (Participants) | 27
Participants | 27

5. Secondary Outcome: Retention Feasibility
Description: Retention feasibility will be measured by calculating the proportion of participants who completed the three month (final) intervention visit out of participants randomized to the intervention arm who completed at least one intervention session..
Time Frame: 3 months
Population: Number of participants randomized to the intervention arm who completed at least 1 intervention session.
Measure: Count of Participants; unit: Participants
Arm/Group | T.A.K.E. Steps Motivational Interviewing Intervention
Number analyzed (Participants) | 42
Participants | 28

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | T.A.K.E. Steps Motivational Interviewing Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT05215262/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT05215262/ICF_001.pdf